CLINICAL TRIAL: NCT00292812
Title: The Clinical Effects of an Infant Formula Supplemented With Various Concentrations of Nucleotides
Brief Title: Clinical Effects of a Nucleotides-Supplemented Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Materna Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sor4123ctil
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-05

CONDITIONS: Nutritional Requirements
Keywords: Infant nutrition; Nucleotides; Infant formula
MeSH Terms: interventions — Dietary Supplements; Nucleotides

INTERVENTIONS:
Drug: Nutritional supplementation (nucleotides)

SUMMARY:
The study hypothesis is that different concentrations of nucleotides' supplementation of an infant formula might affect differently growth and/or other clinical parameters in neonates.

DETAILED DESCRIPTION:
Three groups of 50 newborn infants each, will be fed for 30 days an infant formula supplemented with either 4.9 mg/100 kcal or 10.6 mg/100 kcal of nucleotides or with no supplementation. Newborns will be monitored prospectively for the following outcome parameters:

* Growth percentiles.
* Behaviour and infantile colic.
* Bowel habits.
* Side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns aged 0-30 days.

Exclusion Criteria:

* Prematurity
* Chronic illness
* Failure to thrive
* Milk allergy

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2006-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Growth percentiles, Behaviour and infantile colic, Bowel habits.

SECONDARY OUTCOMES:
Side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Weizman, MD, Principal Investigator — Head, Pediatric GI and Nutrition Unit
Locations (1):
- Soroka Medical Center, Beersheba, Israel